CLINICAL TRIAL: NCT03429166
Title: Connecting Women to Care: Home-based Psychotherapy for Women With MST Living in Rural Areas
Acronym: CWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 16-070
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The current study proposes a blending of design components of clinical effectiveness and implementation research for the purposes increasing translational gains and providing useful information to inform future implementation that would otherwise not be available or take much longer to obtain. This Hybrid Type 1 design combines a randomized clinical effectiveness trial with a mixed-method, multi-stakeholder process evaluation of the delivery of the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STAIR stands for Skills Training in Affective and Interpersonal Regulation (Experimental): STAIR stands for Skills Training in Affective and Interpersonal Regulation a non-trauma-focused treatment
  Interventions: Behavioral: Skills Training in Affective and Interpersonal Regulation
- Present Centered Therapy (Active Comparator): PCT , a non-trauma-focused treatment
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Skills Training in Affective and Interpersonal Regulation — A non-trauma-focused treatment
  Other Names: STAIR
  Arms: STAIR stands for Skills Training in Affective and Interpersonal Regulation
Behavioral: Present Centered Therapy — A non-trauma-focused treatment
  Arms: Present Centered Therapy

SUMMARY:
Military sexual trauma (MST) is a common duty-related stressor which occurs among one in four female Veterans and is associated with substantial concerns about social isolation and high rates of PTSD. Women with MST also experience numerous person-level barriers to care including the desire to avoid male-dominated VA clinics, transportation difficulties and childcare responsibilities. Treatment programs that address the social and mental health needs of this population and acknowledge barriers to care that disproportionately affect women are lacking. The proposed study will use a hybrid effectiveness-implementation design to evaluate the in-home delivery of a gender-sensitive, evidence-based coping skills program to improve social and role functioning as well as reduce PTSD and will prioritize enrolling rural women in a representative manner. If the program is found to be successful at improving social functioning and PTSD, and in reducing barriers to care, it will provide a tremendous benefit to women Veterans with MST, particularly those in rural areas.

DETAILED DESCRIPTION:
Background - Military Sexual Trauma (MST) among women Veterans is a problem of epidemic proportion associated with significant mental health and functional impairment and substantial access to care barriers. Surveillance data indicate that one in four women Veterans reports MST when screened. Compared to women Veterans with other service-related stressors, those experiencing MST have greater mental health problems, are more likely to report difficulty in functioning in social, family and intimate relationships and are more likely to be unemployed and to report difficulties in finding a job. Nevertheless, women with MST engage less frequently in VA health care than other women Veterans. Barriers to care include distance from specialty services, financial difficulties, childcare and family responsibilities, and gender-related discomfort in male-dominated VA facilities. Research over the past decade has identified the problems and concerns of women Veterans with MST but programs addressing their mental health needs and responsive to identified barriers are lacking. The proposed study addresses this gap by evaluating a gender-sensitive, evidence-based skills training program delivered via home-based video technology (HBVT).

Specific Aims - The study will conduct a Hybrid Type 1 effectiveness-implementation study to accomplish two aims. The first is to determine the effectiveness of the HBVT-delivered, Skills Training in Affective Regulation (STAIR) relative to a HBVT-delivered nonspecific active comparator, Present Centered Therapy (PCT) among women Veterans with MST. It is hypothesized that STAIR will be superior to PCT in regards to improvement in PTSD symptoms as measured by the Clinician Administered PTSD Scale (CAPS) (primary outcome) as well as in perceived social support and social engagement (secondary outcomes). The second aim is to conduct a multi-stakeholder, mixed method evaluation to inform future potential implementation plans by identify barriers and facilitators of implementing STAIR via HBVT and to contextualize and interpret the quantitative data on treatment processes and clinical effectiveness.

Methodology - This is a four-year, two-site Hybrid Type 1 effectiveness-implementation study design. A total of 200 women Veterans with MST and PTSD symptoms with cut-off of 3 or more from the Diagnostic Statistical Manual 5 (DSM-5) PTSD Screen will be enrolled into the study. Participants will be stratified by rurality status in a proportion representative of the national population (34% rural vs. 66% nonrural). Stratification will ensure that resources are dedicated to recruit the identified number of rural women. Within each level of stratification, participants will be randomized into one of two treatments conditions, STAIR or PCT, each of which is comprised of 10 weekly sessions. Assessments will be conducted at five time-points: baseline (week 0), mid-treatment (week 8), immediately posttreatment (week 16), 2-month follow-up (week 24) and 4-month follow-up (week 32). Rurality will be included as a covariate and assessed for variations in aspects such as retention and outcome, which will help inform future implementation plans. Multi-stakeholder mixed-method process evaluation concerning STAIR and the use of in-home delivery of services will include administrator, clinician and patient stakeholders.

Expected Results and Anticipated Impacts on Veterans Healthcare - It is expected that the proposed study has the potential to improve the quality of VA healthcare by establishing the effectiveness of a social skills intervention, Skills Training in Affective and Interpersonal Regulation (STAIR) delivered via home-based video technology (HBVT) to women Veterans with MST, particularly those living in rural areas. The treatment simultaneously addresses social concerns and PTSD symptoms, both of which are identified needs of women Veterans who have experienced MST. STAIR has been demonstrated as efficacious in community populations and pilot data with women Veterans with MST indicate similar outcomes regarding improvements in perceived social support, social engagement and PTSD symptoms. The use of HBVT has the potential of increasing access to care to this geographically dispersed and underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* A positive screen for MST
* A positive PTSD screen defined as PC-PTSD cut-off of > 3

Exclusion Criteria:

* Substance abuse not in remission for at least 3 months
* Current psychotic symptoms

  * unmedicated mania or bipolar disorder
  * prominent current suicidal or homicidal ideation
* Cognitive impairment indicated by chart diagnoses or observable cognitive difficulties
* Current involvement in a violent relationship defined as more than casual contact

  * e.g., dating or living with an abusive partner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 204 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylene Cloitre, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss BJ, Azevedo K, Webb K, Gimeno J, Cloitre M. Telemental Health Delivery of Skills Training in Affective and Interpersonal Regulation (STAIR) for Rural Women Veterans Who Have Experienced Military Sexual Trauma. J Trauma Stress. 2018 Aug;31(4):620-625. doi: 10.1002/jts.22305. Epub 2018 Aug 2. PMID 30070399
- [Result] Jackson C, Weiss BJ, Cloitre M. STAIR Group Treatment for Veterans with PTSD: Efficacy and Impact of Gender on Outcome. Mil Med. 2019 Jan 1;184(1-2):e143-e147. doi: 10.1093/milmed/usy164. PMID 30007286
- [Result] Cloitre M, Khan C, Mackintosh MA, Garvert DW, Henn-Haase CM, Falvey EC, Saito J. Emotion regulation mediates the relationship between ACES and physical and mental health. Psychol Trauma. 2019 Jan;11(1):82-89. doi: 10.1037/tra0000374. Epub 2018 May 10. PMID 29745688
- [Result] Ben-Ezra M, Karatzias T, Hyland P, Brewin CR, Cloitre M, Bisson JI, Roberts NP, Lueger-Schuster B, Shevlin M. Posttraumatic stress disorder (PTSD) and complex PTSD (CPTSD) as per ICD-11 proposals: A population study in Israel. Depress Anxiety. 2018 Mar;35(3):264-274. doi: 10.1002/da.22723. Epub 2018 Feb 16. PMID 29451956
- [Result] Schnyder U, Schafer I, Aakvaag HF, Ajdukovic D, Bakker A, Bisson JI, Brewer D, Cloitre M, Dyb GA, Frewen P, Lanza J, Le Brocque R, Lueger-Schuster B, Mwiti GK, Oe M, Rosner R, Schellong J, Shigemura J, Wu K, Olff M. The global collaboration on traumatic stress. Eur J Psychotraumatol. 2017 Nov 30;8(sup7):1403257. doi: 10.1080/20008198.2017.1403257. eCollection 2017. PMID 29435201
- [Result] Cloitre M, Garvert DW, Weiss BJ. Depression as a moderator of STAIR Narrative Therapy for women with post-traumatic stress disorder related to childhood abuse. Eur J Psychotraumatol. 2017 Oct 10;8(1):1377028. doi: 10.1080/20008198.2017.1377028. eCollection 2017. PMID 29038682
- [Result] Hyland P, Shevlin M, Cloitre M, Karatzias T, Vallieres F, McGinty G, Fox R, Power JM. Quality not quantity: loneliness subtypes, psychological trauma, and mental health in the US adult population. Soc Psychiatry Psychiatr Epidemiol. 2019 Sep;54(9):1089-1099. doi: 10.1007/s00127-018-1597-8. Epub 2018 Oct 6. PMID 30293176
- [Result] Karatzias T, Hyland P, Bradley A, Fyvie C, Logan K, Easton P, Thomas J, Philips S, Bisson JI, Roberts NP, Cloitre M, Shevlin M. Is Self-Compassion a Worthwhile Therapeutic Target for ICD-11 Complex PTSD (CPTSD)? Behav Cogn Psychother. 2019 May;47(3):257-269. doi: 10.1017/S1352465818000577. Epub 2018 Oct 2. PMID 30277191
- [Result] Kazlauskas E, Gegieckaite G, Hyland P, Zelviene P, Cloitre M. The structure of ICD-11 PTSD and complex PTSD in Lithuanian mental health services. Eur J Psychotraumatol. 2018 Jan 11;9(1):1414559. doi: 10.1080/20008198.2017.1414559. PMID 33680347
- [Result] Olff M, Amstadter A, Armour C, Birkeland MS, Bui E, Cloitre M, Ehlers A, Ford JD, Greene T, Hansen M, Lanius R, Roberts N, Rosner R, Thoresen S. A decennial review of psychotraumatology: what did we learn and where are we going? Eur J Psychotraumatol. 2019 Nov 20;10(1):1672948. doi: 10.1080/20008198.2019.1672948. eCollection 2019. PMID 31897268
- [Result] Coventry PA, Meader N, Melton H, Temple M, Dale H, Wright K, Cloitre M, Karatzias T, Bisson J, Roberts NP, Brown JVE, Barbui C, Churchill R, Lovell K, McMillan D, Gilbody S. Psychological and pharmacological interventions for posttraumatic stress disorder and comorbid mental health problems following complex traumatic events: Systematic review and component network meta-analysis. PLoS Med. 2020 Aug 19;17(8):e1003262. doi: 10.1371/journal.pmed.1003262. eCollection 2020 Aug. PMID 32813696
- [Result] Ho GWK, Karatzias T, Vallieres F, Bondjers K, Shevlin M, Cloitre M, Ben-Ezra M, Bisson JI, Roberts NP, Astill Wright L, Hyland P. Complex PTSD symptoms mediate the association between childhood trauma and physical health problems. J Psychosom Res. 2021 Mar;142:110358. doi: 10.1016/j.jpsychores.2021.110358. Epub 2021 Jan 12. PMID 33508705
- [Result] McGinty G, Fox R, Ben-Ezra M, Cloitre M, Karatzias T, Shevlin M, Hyland P. Sex and age differences in ICD-11 PTSD and complex PTSD: An analysis of four general population samples. Eur Psychiatry. 2021 Oct 4;64(1):e66. doi: 10.1192/j.eurpsy.2021.2239. PMID 34602122
- [Derived] Rashkovsky K, Morabito DM, Chargin B, Chang CJ, Morland LA, Cloitre M. Treatment outcomes of sexual minority women (SMW) veterans with military sexual trauma (MST). Psychol Trauma. 2025 Dec 18:10.1037/tra0002077. doi: 10.1037/tra0002077. Online ahead of print. PMID 41411035
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 305 candidates who completed screens, 204 completed baseline and 161 met study criteria and were randomized.
Period: Overall Study
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Started | 79 | 82
Completed | 66 | 70
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Present Centered Therapy: Present Centered Therapy (PCT) a non-trauma-focused treatment
  Present Centered Therapy: A non-trauma-focused treatment
- Total: Total of all reporting groups
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy | Total
Number analyzed (Participants) | 79 | 82 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 82 | 161
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 82 | 161
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 6 | 15
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 17 | 17 | 34
  White | 45 | 48 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 82 | 161
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity [Mean (Standard Deviation); unit: units on a scale] — (CAPS-5) Total Severity score range of 0 to 80 where higher is worse.
  units on a scale | 41.74 (11.88) | 43.06 (11.43) | 42.41 (11.70)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessed Severity of PTSD
Description: Clinician Administered PTSD Scale for the Diagnostic Statistical Manual Fifth Edition (DSM-5) (CAPS-5) Total Severity CAPS-5 is a clinician administered interview which assesses DSM-5 symptom severity and diagnosis. The measure includes 20 items rated on a 5-point Likert scale which ranges from 0 to 80 where higher scores mean worse outcomes.
Time Frame: Baseline, 16, 24 and 32 weeks
Population: Intent to Treat Analysis is complete for 16 weeks (immediately posttreatment) and 24 weeks (2 month follow-up) and 32 weeks (4 month follow-up)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 41.74 (11.88) | 43.06 (11.43)
  Post-treatment (week 16) | 27.78 (7.69) | 34.00 (7.47)
  2-Month Follow-Up (week 24) | 28.88 (7.87) | 34.05 (7.64)
  4-Month Follow-Up (week 32) | 29.98 (7.87) | 34.10 (7.64)

2. Secondary Outcome: PTSD Symptom Severity (Self-Report)
Description: PTSD Checklist for DSM-5 (PCL-5) is a 20 item measure with a Likert scale from 0 to 4. Possible total scores range from 0 to 80, where higher scores indicate more severe symptoms.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 47.52 (7.43) | 49.12 (7.23)
  Midtreatment (week 8) | 38.17 (9.09) | 41.88 (8.80)
  Posttreatment (week 16) | 28.82 (9.09) | 34.64 (8.80)
  2-month Follow-Up (week 24) | 30.36 (9.20) | 36.57 (8.89)
  4-month Follow-up (week 32) | 31.90 (9.20) | 38.49 (8.89)

3. Secondary Outcome: Social Support
Description: Interpersonal Support Evaluation List -12 (ISEL-12) is a 12 item measure of social support with a Likert scale from 0 to 3. Possible total scores range from 0 to 120 with higher scores indicate greater perceived support.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 68.16 (9.81) | 65.49 (9.55)
  Midtreatment (week 8) | 72.30 (11.77) | 66.92 (11.42)
  Posttreatment (week 16) | 76.44 (11.77) | 68.34 (11.42)
  2-Month Follow-Up (week 24) | 74.65 (11.90) | 68.01 (11.52)
  4-Month Follow-Up (week 32) | 72.86 (11.90) | 67.67 (11.52)

4. Secondary Outcome: Emotion Regulation Difficulties
Description: Difficulties in Emotion Regulation Scale-36 (DERS-36) is a 36 item self-report measure of emotion regulation difficulties that is rated on a scoe of 0 to 5. Possible total scores range from 0 to 180 where higher scores indicate more difficulties.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 107.31 (9.92) | 109.51 (9.37)
  Midtreatment (week 8) | 96.79 (11.95) | 103.48 (11.61)
  Posttreatment (week 16) | 86.26 (11.95) | 97.45 (11.61)
  2-Month Follow-Up (week 24) | 85.67 (12.14) | 97.63 (11.76)
  4-Month Follow-Up (week 32) | 85.07 (12.14) | 97.80 (11.76)

5. Secondary Outcome: Depression
Description: Beck Depression Inventory-11 (BDI-11) is an 11 item measure. Possible total scores can range from 0 to 63 where higher scores mean more depression.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 35.50 (4.97) | 36.13 (4.84)
  Midtreatment (week 8) | 29.27 (6.14) | 32.10 (5.95)
  Posttreatment (week 16) | 23.04 (6.14) | 28.06 (5.95)
  2-Month Follow-Up (Week 24) | 23.78 (6.24) | 28.37 (6.03)
  4-Month Follow-Up (week 32) | 24.51 (6.24) | 28.67 (6.03)

6. Secondary Outcome: Posttraumatic Maladaptive Beliefs
Description: Posttraumatic Maladaptive Belief Scale (PMBS) is a 15 item self-report measure. Responses are measured on a 7-point scale from 0 to 6. Possible total scores range from 0 to 90 where higher scored indicate strong maladaptive beliefs.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 46.73 (13.15) | 48.44 (14.56)
  Midtreatment (week 8) | 41.79 (7.72) | 45.99 (7.49)
  Posttreatment (week 16) | 36.74 (7.72) | 43.01 (7.49)
  2-Month Follow-Up (week 24) | 37.47 (7.80) | 42.87 (7.55)
  4-Month Follow-Up (week 32) | 38.19 (7.80) | 42.73 (7.55)

7. Secondary Outcome: Psychosocial Functioning
Description: The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) Life Activities Subscale is an 8 item measure of how difficult daily life activities are to complete. Responses range from 0 to 4. Possible total scores range from 0 to 32 with higher scores indicating greater difficulties.
Time Frame: Baseline, 8, 16, 24 and 32 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
Number analyzed (Participants) | 79 | 82
score on a scale
  Baseline (week 0) | 14.88 (3.48) | 15.10 (3.39)
  Midtreatment (week 8) | 13.07 (4.31) | 13.47 (4.18)
  Posttreatment (week 16) | 11.26 (4.31) | 11.84 (4.18)
  2-Month Follow-Up (week 24) | 11.61 (4.37) | 12.32 (4.23)
  4-Month Follow-Up (week 32) | 11.96 (4.37) | 12.80 (4.23)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs), Adverse Events (AEs) and deaths were collected from the time of study entry until the end of study participation including treatment follow-up, an average of 32 weeks.
Arm/Group | STAIR Stands for Skills Training in Affective and Interpersonal Regulation | Present Centered Therapy
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/82
Other Adverse Events (participants affected / at risk) | 0/79 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03429166/Prot_SAP_000.pdf